CLINICAL TRIAL: NCT04609254
Title: Comparison of The Effectiveness of Intravenous Paracetamol, Dexketoprofen and Ibuprofen In The Treatment of Non-Traumatic Acute Low Back Pain In The Emergency Department
Brief Title: Paracetamol, Dexketoprofen and Ibuprofen In Non-Traumatic Acute Low Back Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Ibrahim Turkcuer, Professor, MD, Pamukkale University
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: 2019TIPF007
Record Dates: First submitted 2020-10-26; First posted 2020-10-30 (Actual); Last update posted 2020-10-30 (Actual); Status verified 2020-10

CONDITIONS: Low Back Pain, Mechanical
Keywords: paracetamol; dexketoprofen; ibuprofen; emergency department; low back pain
MeSH Terms: conditions — Low Back Pain; Emergencies | interventions — Acetaminophen; dexketoprofen trometamol; Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- First Group (Experimental): 1000 mg of paracetamol ( parol 1000mg vial-atabay chemistry-İstanbul) intravenous (IV) was given 71 patients,
  Interventions: Drug: Paracetamol
- Second Group (Experimental): dexketoprofen 50 mg arveles 50 mg ampoule -Menarini- Istanbul) intravenous (IV) was given 70 patients,
  Interventions: Drug: Dexketoprofen
- Third group (Experimental): 400 mg Ibuprofen (İntrafen 400 mg vial- Gen-İstanbul) intravenous (IV) was given 69 patients, which determined to be applied as a group.
  Interventions: Drug: Ibuprofen

INTERVENTIONS:
Drug: Paracetamol — 1000 mg of paracetamol ( parol 1000mg vial-atabay chemistry-İstanbul) intravenous (IV) was given 71 patients,
  Other Names: Perfalgan
  Arms: First Group
Drug: Dexketoprofen — dexketoprofen 50 mg arveles 50 mg ampoule -Menarini- Istanbul) intravenous (IV) was given 70 patients,
  Other Names: ASEKET; DARKIN; DEXALGIN; DESTIYO; DEXCORIL
  Arms: Second Group
Drug: Ibuprofen — 400 mg Ibuprofen (İntrafen 400 mg vial- Gen-İstanbul) intravenous (IV) was given 69 patients, which determined to be applied as a group.
  Other Names: İntrafen
  Arms: Third group

SUMMARY:
* Currently, paracetamol and nonsteroidal antiinflammatory drugs are widely used by emergency physicians in Turkey for the treatment of patients with Non-Traumatic Acute Low Back Pain
* The objective of the study is compare the efficacy of intravenous dexketoprofen,ibuprofen with paracetamol in the treatment of Non-Traumatic Acute Low Back Pain

DETAILED DESCRIPTION:
* This is the randomized double blinded clinical trial to compare the efficacy of these three drugs in this clinical setting.
* A randomized clinical trial was conducted in the Emergency Department (ED) of Pamukkale University Medical Faculty Hospital
* Study personnel (emergency physicians and nurses) were trained before the study.
* When intravenous drugs (Paracetamol, Dexketoprofen and ibuprofen) was being recommended, an eligibility checklist was completed by the attending physician.
* If there were no exclusion criteria, written informed consent was obtained and baseline information, including initial Non-Traumatic Acute Low Back Pain severity ratings with visual analog scale (VAS) were recorded.
* The need for identification and enrollment of participants by staff with conflicting work pressures resulted in recruitment of a convenience sample of patients.
* All patients eligible for the study were randomized to one of three groups:

First Group: 1000 mg of paracetamol (parol 1000mg vial-atabay chemistry-İstanbul ) intravenous (IV) was given 71 patients, Second Group: dexketoprofen 50 mg ( arveles 50 mg ampoule -Menarini- Istanbul) intravenous (IV) was given 70 patients, third group: 400 mg İbuprofen (İntrafen 400 mg vial- Gen-İstanbul) intravenous (IV) was given 69 patients, which determined to be applied as a group. Drug packs prepared in 150 ml serum physiology were numbered by an independent nurse, who not involved in the study.

* Drugs were prepared according to the computer-generated random number sequence to assign treatment allocations
* The allocation list was kept by the emergency nurse. Patients received the paracetamol,dexketoprofen,ibuprofen medication schemes according to their random allocations.
* After enrollment and recording of baseline information, the next numbered study drug pack was obtained, and administered intravenously.
* Randomization was achieved by using computer software to generate random numbers. During the intervention, participants were monitored by an oxygen saturation (SpO2) monitor, an automatic sphygmomanometer (blood pressure), and a rhythm monitor (heart rate and rhythms)
* One researcher blinded to patient allocation observed the whole procedure and recorded the Non-Traumatic Acute Low Back Pain scores.
* Patients in three groups received three types of medication in a similar manner, thus ensuring double blind.

Non-Traumatic Acute Low Back Pain scores were recorded at 0, 15, 30 and 60 min on a VAS of 1 to 100

• During the study, pulse rate, systolic blood pressure, diastolic blood pressure, respiration rate and oxygen saturation (SpO2) were recorded at baseline (0 min), 15, 30, and 60 min.

ELIGIBILITY:
Inclusion Criteria:

* • Patients were eligible for inclusion if they were aged 18 years or older, 65 years or younger Isolated non traumatic musculoskeletal pain Patients who agree to work and receive the approval VAS (visual analog scale) score>5.

Exclusion Criteria:

* • Patients with severe liver, kidney,pulmonary and cardiac heartfailure

  * To be Pregnancy and breast-feeding
  * Have received analgesics in the last 6hours
  * Patients of childbearing age who are not using a birth control method.
  * Patients with neurological deficits
  * Patients with cardiac chest pain
  * Patients with chronic pain
  * Patients with pre-existing ibuprofen, dexketoprofen and paracetamolinduced gastrointestinal bleeding and perforation
  * Patients with reflected pain
  * Patients with neoplastic pain
  * Patients with an allergy trait (ibuprofen, paracetamol and dexketoprofen)
  * Illiterates and patients with vision problems

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2018-12-15 (Actual); Primary Completion 2020-04-15 (Actual); Study Completion 2020-09-15 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in Non-Traumatic Acute Low Back Pain on the Visual Analog Scale at 60 minutes | Baseline and 60 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Cansu Dogan, MD, Principal Investigator — Pamukkale University
Locations (1):
- Pamukkale University, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will be made available to other researchers whenever they need it.